CLINICAL TRIAL: NCT04284644
Title: A Novel Co-induction Technique Compared to Standard Inhalational and Intravenous Induction Techniques: a Prospective Randomized Control Study
Brief Title: Co-induction Technique Compared to Standard Inhalational and Intravenous Induction Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, omar ahmad ababneh, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10/2016/4597
Record Dates: First submitted 2020-02-20; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia; Anesthesia; Adverse Effect
Keywords: General anesthesia; Propofol; Sevoflurane; Co-induction; Laryngeal mask airway
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group P (Experimental): Patient received a dose of 1.5 mg/kg of Propofol slowly over 2 minutes for induction.
  Interventions: Drug: Induction using propofol
- Group S (Experimental): Patient received 8% sevoflurane through sealed plastic facemask at 8 L/min flow of oxygen.
  Interventions: Drug: Induction using sevoflurane
- Group C (Experimental): Patient received 4% sevoflurane through sealed plastic facemask at 8 L/min flow of oxygen for 2 minutes, followed by a dose of 0.75 mg/kg of propofol given slowly.
  Interventions: Drug: Induction using propofol and sevoflurane

INTERVENTIONS:
Drug: Induction using propofol — Patients were given 1.5 mcg/Kg of fentanyl intravenously. two minutes after the fentanyl dose, a dose of 1.5 mg/kg of propofol slowly over 2 minutes.
  Arms: Group P
Drug: Induction using sevoflurane — Patients were given 1.5 mcg/Kg of fentanyl intravenously. two minutes after the fentanyl dose, patient received 8% inhalational sevoflurane through sealed plastic face mask at 8 L/min flow of oxygen.
  Arms: Group S
Drug: Induction using propofol and sevoflurane — Patients were given 1.5 mcg/Kg of fentanyl intravenously. two minutes after the fentanyl dose, patient received 4% sevoflurane through sealed plastic face mask at 8 L/min flow of oxygen for 2 minutes, followed by a dose of 0.75 mg/kg of propofol given slowly.
  Arms: Group C

SUMMARY:
Co-induction technique refers to the use of a combination of medications to reach the desired therapeutic target. In the present study, the investigators examined the safety of a novel co-induction approach that relied on a simple timing and dosing alterations to the classical approaches of inhalational sevoflurane and propofol induction. The significance of this study is to find a reliable safe alternative method of induction that can provide optimal parameters,when compared to the classical methods of induction.

DETAILED DESCRIPTION:
Co-induction technique refers to the use of a combination of medications to reach the desired therapeutic target. This technique is considered an approach that can be of a great benefit to patients with chronic medical illnesses and those who have moderate to high risk for general anaesthesia.

In the present study, the investigators examined the safety of a novel co-induction approach that relied on a simple timing and dosing alterations to the classical approaches of inhalational sevoflurane and propofol induction. The significance of this study is to find a reliable safe alternative method of induction that can provide optimal parameters,when compared to the classical methods of induction. The investigators evaluated the time needed for laryngeal mask airway (LMA) insertion, number of LMA insertion trials, succession of LMA insertion, adverse events related to the airway, respiratory and cardiovascular systems, haemodynamic stability and satisfaction scores of enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with Age ≥ 65 years.
* American Society of Anaesthesiologists' (ASA) score II or III.
* minimally invasive endoscopic urological procedures.

Exclusion Criteria:

* patient refusal.
* Age < 65 years.
* family history of malignant hyperthermia.
* prolonged surgery that needed intubation.
* body mass index (BMI) > 35 kg/m2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
Intraoperative respiratory adverse events | 8 months
  The investigators recorded the occurrence of transient apnea intraoperatively, in addition to laryngeal spasm, coughing, gagging and increased salivation. The study chart included the documentation these common adverse events, the timing of occurrence, and the intervention required to manage these events.

SECONDARY OUTCOMES:
Time for successful laryngeal mask airway insertion | 8 months
  The investigators assessed the time needed for LMA insertion. The timer was started upon giving the fentanyl, recording the time till successful insertion of laryngeal mask airway.
Blood pressure stability | 8 months
  The investigators recorded patients' blood pressure readings throughout the induction procedure.
Heart rate stability | 8 months
  The investigators recorded patients' heart rate throughout the induction procedure.
Changes in oxygen saturation | 8 months
  The investigators recorded patients' oxygen saturation throughout the induction procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No